CLINICAL TRIAL: NCT03568227
Title: Multimodal Investigation of Distinct Hypnotic States - A Resting-State fMRI Study
Brief Title: Hemodynamic Correlates of Distinct Hypnotic States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike Bruegger (Other)
Responsible Party: Sponsor-Investigator, Mike Bruegger, Senior Researcher, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HypnoScienceMRI
Record Dates: First submitted 2018-06-07; First posted 2018-06-26 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Hypnosis
Keywords: Hypnosis; Neurophysiology; fMRI; Resting-State; Hypnotic Sub-States
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): The study has a 2 (Intervention: Hypnosis, Control) x 2 (State: 1 & 2) factorial within-subjects design, resulting in a total of 4 conditions. All volunteers participate at the 4 conditions in the same session.The order of the interventions is counterbalanced resulting in two possible sequences:
  Sequence 1: Hypnosis State 1, Hypnosis State 2, Control State 1, Control State 2
  Sequence 2: Control State 1, Control State2, Hypnosis State 1, Hypnosis State 2
  Volunteers will be randomly allocated to the two sequence types.
  Interventions: Procedure: Hypnosis; Procedure: Control

INTERVENTIONS:
Procedure: Hypnosis — The hypnosis intervention consists of two elements: A hypnotic induction and a hypnotic deepening. The induction aims at guiding the participant into the first hypnotic state (state 1). The participants will remain in this state for 10 minutes, the duration of the fMRI-scan. The hypnotic deepening guides the participants into a very deep hypnotic state (state 2). Participants also remain in this state for 10 minutes, during which their brain activity is measured using fMRI
Procedure: Control — The control intervention consists of texts corresponding to the induction and deepening of the hypnosis intervention. They are matched in duration and consist of textually matched excerpts from www.wikipedia.org. Control induction will be presented, resulting in the control state 1 (10 min). Then the control deepening will be performed, leading to the control state 2 (10 minutes). During both control states the brain activity will be recorded using fMRI.

SUMMARY:
The investigation will assess the brain activation connectivity patterns associated with hypnosis and possible hypnotic sub-states by means of functional magnetic resonance imaging (fMRI). For that purpose, 50 healthy participants highly familiar with hypnosis (according to the OMNI-method) will be recruited and tested.

DETAILED DESCRIPTION:
Despite the growing number of studies investigating of the physiological underpinnings of hypnosis by means of neuroimaging methods such as electroencephalography (EEG) positron emission tomography (PET) and functional magnetic resonance imaging (fMRI), still no consensus exists regarding the underlying neurophysiological working mechanisms due to high levels of variability in the data.

Generally, the variability observed in research examining the neurobiological fundamentals of hypnosis could be attributed to the following characteristics:

1. Heterogeneity regarding hypnotic induction procedures.
2. Insufficient statistical power.
3. Mono-Modality: Studies investigating the neurophysiologic mechanisms of hypnosis typically apply only one method for the investigation of their research questions. However, different techniques complement each other, hence, resulting in a more thorough understanding of the mechanisms of action.

In this project, the investigators present a multimodal approach, in which these three points are considered in order to provide a comprehensive picture with respect to psycho- and neurophysiologic fundamentals of hypnosis and proposed distinct hypnotic states.

Point 1) will be approached by applying a highly reproducible method for the hypnotic induction (OMNI-hypnosis). This hypnosis method is fast, direct and all OMNI educated hypnotherapists follow exactly the same induction procedure. This implies a high level of standardization and operationalization, crucial prerequisites to investigate the phenomenon based on scientific guidelines.

Point 2) will be addressed by including a homogeneous study sample of 50 highly suggestible participants. Furthermore, the comparably high number of 50 participants should ensure sufficient statistical power particularly in consideration of the homogeneity of the study sample.

Point 3) is addressed by following a multimodal approach combining a vast array of psychophysiological measures with multimodal neuroimaging. For that purpose, the project will be divided into three studies: A EEG- and psychophysiological study, a fMRI-study and a magnetic resonance spectroscopy (1H-MRS) study.

In the present study, fMRI is applied for the investigation of network dynamics associated with hypnotic states. Hypnotic states will be compared to control states which follow mock instructions matched to the hypnosis instructions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65
* Proficient in German language
* Written informed consent after being informed
* Familiar with hypnotic states of OMNI-Hypnosis

Exclusion Criteria:

* Pre-existing neurological and/or psychiatric conditions
* History of brain injuries
* Alcohol and/or drug abuse
* Chronic diseases that require a permanent intake of drugs

Additional exclusion criteria for the MRI- and 1H-MRS-experiment:

* General contraindications for a participation on a MRI-Experiment (e.g. claustrophobia, pace maker, cochlea implants, insulin pumps)
* Hypersensitivity to loud noise
* Not being able to lie still during a longer period of time
* Foreign metallic objects in the body (e.g. gunshot wounds, metallic particles, metal implants, irremovable piercings)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Differences in resting state functional connectivity (assessed using fMRI) between the four conditions (control state 1 & 2, hypnotic state 1 & 2) | 90 minutes

SECONDARY OUTCOMES:
Differences in heart rate variability (assessed during fMRI measurements) between the four conditions (control state 1 & 2, hypnotic state 1 & 2) | 90 minutes
Differences respiratory frequency (assessed during fMRI measurements) between the four conditions (control state 1 & 2, hypnotic state 1 & 2) | 90 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Elkins GR, Barabasz AF, Council JR, Spiegel D. Advancing research and practice: the revised APA Division 30 definition of hypnosis. Int J Clin Exp Hypn. 2015;63(1):1-9. doi: 10.1080/00207144.2014.961870. PMID 25365125
- [Background] Jensen MP, Jamieson GA, Lutz A, Mazzoni G, McGeown WJ, Santarcangelo EL, Demertzi A, De Pascalis V, Banyai EI, Rominger C, Vuilleumier P, Faymonville ME, Terhune DB. New directions in hypnosis research: strategies for advancing the cognitive and clinical neuroscience of hypnosis. Neurosci Conscious. 2017;3(1):nix004. doi: 10.1093/nc/nix004. Epub 2017 Apr 12. PMID 29034102
- [Background] McGeown WJ, Mazzoni G, Vannucci M, Venneri A. Structural and functional correlates of hypnotic depth and suggestibility. Psychiatry Res. 2015 Feb 28;231(2):151-9. doi: 10.1016/j.pscychresns.2014.11.015. Epub 2014 Dec 6. PMID 25557062
- [Background] Terhune DB, Cleeremans A, Raz A, Lynn SJ. Hypnosis and top-down regulation of consciousness. Neurosci Biobehav Rev. 2017 Oct;81(Pt A):59-74. doi: 10.1016/j.neubiorev.2017.02.002. Epub 2017 Feb 4. PMID 28174078
- [Background] Varga K, Kekecs Z, Myhre PS, Jozsa E. A Neutral Control Condition for Hypnosis Experiments: "Wiki" Text. Int J Clin Exp Hypn. 2017 Oct-Dec;65(4):429-451. doi: 10.1080/00207144.2017.1348833. PMID 28836922